CLINICAL TRIAL: NCT05508295
Title: Setting up a Community Based Patient Cohort to Understand Long COVID: Monoclonal Antibody and Post-Infection COVID Vaccine Administration as the FOCI
Brief Title: Long COVID-19 and MAB Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MultiCare Health System Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 02/01/2022
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID positive case with mAb treatment
- COVID positive case having not received mAb treatment
- COVID negative cases

SUMMARY:
This study will be observational only. It will provide real-world evidence generated from a representative and large-scale COVID patient base. The adoption, pilot testing and use of NIH PROs among viral tested patients with research purpose on long COVID will be unique and innovative. With the existing and proven scientific rigor, NIH PRO system will be adopted, then modified and tailored to form the long hauler specific, comprehensive instrument, helping generalize future knowledge regarding COVID-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Have been tested for COVID at one of the MultiCare facilities,
* AND 18 years old or older at the viral test,
* AND have no problem understanding English or Spanish.

Exclusion Criteria:

* Pediatric patients younger than 18 years old at the time of testing,
* OR patients who are pregnant,
* OR patients who plan to get pregnant in 3 months,
* OR patients who are hospitalized at the time of recruitment,
* OR patients who have cognitive impairment(s) at the recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A small representative sample of up to 50 patients (25 hospitalized and alive at the time of the extraction) will be randomly selected and invited to test for the PRO instrument
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Adopt the NIH PROMIS system (The Assessment Center Instrument Library, which includes all Fixed Length Short Form and Computer Adaptive Test/Item Bank instruments from PROMIS) to construct a modified comprehensive PRO instrument. | 18-month study length, with a pilot reliability study.
  Using a modified NIH PRO measurement system. This system will involve different domains and instruments. Patients will answer PRO questions at the time of recruitment (baseline), then followed up 3 months and 6 months after the first survey (follow-up).
  The modified comprehensive PRO instrument will specifically ask patients to report symptoms based on their health status within a fixed time window, and at the time when the survey questions are given.

SECONDARY OUTCOMES:
Selected comorbidities, all-cause hospitalization and ER visits. | 3 months and 6 months follow-up.
  Extracted from patients' electronic health records.
Patients' COVID vaccination and mAb therapy history will be verified based on self report and EHR. | 18-month study length

CONTACTS AND LOCATIONS:
Locations (1):
- MultiCare Health System, Tacoma, Washington, United States